CLINICAL TRIAL: NCT02473107
Title: CARies DEtection in Children - Cost-efficacy, Applicability and Impact on Quality of Life of Detecting Active Initial Caries Lesions in Primary Teeth
Brief Title: Impact of Detecting Initial and Active Caries Lesions in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Mariana Minatel Braga, PhD, Senior Lecturer, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CARDEC-02
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
Keywords: Dental caries; Primary tooth; Caries Detection
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Caries Detection Strategy (Other): Detection and treatment based on more advanced lesions, despite activity status - Advanced caries lesions detection (no activity assessment)
  Interventions: Other: Advanced caries lesions detection (no activity assessment)
- Test Caries Detection Strategy (Other): Detection and treatment based on all detected caries lesions, considering their activity status as a differential in clinical decision-making - All caries lesions detection (+activity assessment)
  Interventions: Other: All caries lesions detection (+activity assessment)

INTERVENTIONS:
Other: Advanced caries lesions detection (no activity assessment) — The diagnosis strategy will based on detection of only moderate and advanced caries lesions (ICDAS scores 3 to 6). Initial caries lesions will be considered as sound surfaces. Caries activity status will not be evaluated. Clinical decision-making will be proposed for all lesions detected, based on evidence-based protocols.
  Other Names: WHO criteria; Advanced caries lesions; Extensive Decays
  Arms: Control Caries Detection Strategy
Other: All caries lesions detection (+activity assessment) — The diagnosis strategy will based on detection of initial, moderate and advanced caries lesions (ICDAS scores 1 to 6). Caries activity status will be also evaluated. Clinical decision-making will be proposed for all active lesions detected, based on evidence-based protocols. inactive caries lesions will not be treated.
  Other Names: Caries activity assessment; initial caries lesions; early detection
  Arms: Test Caries Detection Strategy

SUMMARY:
The present study aims to evaluate the impact of detecting active initial caries lesions in primary teeth regarding effectiveness, cost-effectiveness, applicability (acceptability and satisfaction) and quality of life. For this, 248 children 3-6 years with complete primary dentition will be examined and treated in a mobile dental unit, which will temporarily be parked in public schools of Sao Paulo. The caries detection will be conducted using the International Caries Detection and Assessment System (ICDAS) and, depending on allocation, an adjunct criterion for caries activity assessment. Children will be randomized in two groups according to the caries threshold to be detected: Group A (only advanced lesions will be detected and treated, independently of their activity status) and Group B (all caries lesions, including initial ones, will be detected and all active lesions will be treated). After this, the treatment plan for each child will be made according to strategies mentioned above. Data concerning the cost-effectiveness of the procedures, acceptability / satisfaction of children and quality of life will be collected after diagnosis, after the end of treatment and 12 and 24 months from the initial examination. For comparison between groups, multilevel regression analyses will be performed. The primary outcome will be sites which need of operative treatment during the follow-up periods and the secondary outcomes will be the cost-effectiveness of each strategy, the acceptability / satisfaction of the child and the impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 36 months to 83 months;
* Should have complete primary dentition;
* Children must assent to participate and their parents must consent to their participation by signing the consent form.

Exclusion Criteria:

* Medical and/or behavioral conditions that requires special considerations regarding management/treatment of the child;
* Children involved in other research that may impact on this study;
* Families who are expected to move out of the coverage area of study during the first year of enrollment.

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Incremental number of dental surfaces with operative treatment needs | After 12 and 24 months from allocation
  This outcome will be assessed by the new caries lesions and / or progression of lesions previously diagnosed / treated and number of treated surfaces which will need restoration replacement, endodontic treatment or extraction after the initial treatment.

SECONDARY OUTCOMES:
Cost-efficacy | After 12 and 24 months from the allocation
  The costs of the diagnostic strategy will be calculated and compared with threshold values for intervention cost-effectiveness by region, determined by World Health Organization.
Discomfort | immediately after the allocation and after 12 and 24 months
  Participants' discomfort, measured by a validated scale (Wong-Baker scale).
Impact of oral health on quality of life | 12 and 24 months after the allocation
  Impact of oral health on quality of life of the children participants in the study, measured by a validated questionnaire (ECOHIS).

OTHER OUTCOMES:
Costs | Immediately after allocation
  The costs of each diagnostic strategy and treatment based on that will be calculated, regarding time of each clinical session, materials used, duration of treatment and possible repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, Principal Investigator — University of Sao Paulo; Isabela Floriano, Principal Investigator — University of Sao Paulo; Fausto M Mendes, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Nyvad B, Fejerskov O. Assessing the stage of caries lesion activity on the basis of clinical and microbiological examination. Community Dent Oral Epidemiol. 1997 Feb;25(1):69-75. doi: 10.1111/j.1600-0528.1997.tb00901.x. PMID 9088694
- [Background] Nyvad B. Diagnosis versus detection of caries. Caries Res. 2004 May-Jun;38(3):192-8. doi: 10.1159/000077754. PMID 15153688
- [Background] Baelum V, Heidmann J, Nyvad B. Dental caries paradigms in diagnosis and diagnostic research. Eur J Oral Sci. 2006 Aug;114(4):263-77. doi: 10.1111/j.1600-0722.2006.00383.x. PMID 16911097
- [Background] Ismail AI. Clinical diagnosis of precavitated carious lesions. Community Dent Oral Epidemiol. 1997 Feb;25(1):13-23. doi: 10.1111/j.1600-0528.1997.tb00895.x. PMID 9088688
- [Background] Pitts NB. Are we ready to move from operative to non-operative/preventive treatment of dental caries in clinical practice? Caries Res. 2004 May-Jun;38(3):294-304. doi: 10.1159/000077769. PMID 15153703
- [Background] Ekstrand KR. Improving clinical visual detection--potential for caries clinical trials. J Dent Res. 2004;83 Spec No C:C67-71. doi: 10.1177/154405910408301s13. PMID 15286125
- [Background] Kidd E, Fejerskov O. Changing concepts in cariology: forty years on. Dent Update. 2013 May;40(4):277-8, 280-2, 285-6. doi: 10.12968/denu.2013.40.4.277. PMID 23829008
- [Background] Baelum V, Machiulskiene V, Nyvad B, Richards A, Vaeth M. Application of survival analysis to carious lesion transitions in intervention trials. Community Dent Oral Epidemiol. 2003 Aug;31(4):252-60. doi: 10.1034/j.1600-0528.2003.00045.x. PMID 12846847
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Piovesan C, Ardenghi TM, Guedes RS, Ekstrand KR, Braga MM, Mendes FM. Activity assessment has little impact on caries parameters reduction in epidemiological surveys with preschool children. Community Dent Oral Epidemiol. 2013 Jun;41(3):204-11. doi: 10.1111/cdoe.12004. Epub 2012 Sep 25. PMID 23004568
- [Background] Mendes FM, Braga MM, Oliveira LB, Antunes JL, Ardenghi TM, Bonecker M. Discriminant validity of the International Caries Detection and Assessment System (ICDAS) and comparability with World Health Organization criteria in a cross-sectional study. Community Dent Oral Epidemiol. 2010 Oct;38(5):398-407. doi: 10.1111/j.1600-0528.2010.00557.x. PMID 20636415
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Background] Harris R, Gamboa A, Dailey Y, Ashcroft A. One-to-one dietary interventions undertaken in a dental setting to change dietary behaviour. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006540. doi: 10.1002/14651858.CD006540.pub2. PMID 22419315
- [Background] Liu BY, Lo EC, Chu CH, Lin HC. Randomized trial on fluorides and sealants for fissure caries prevention. J Dent Res. 2012 Aug;91(8):753-8. doi: 10.1177/0022034512452278. Epub 2012 Jun 26. PMID 22736448
- [Background] Ricketts DN, Kidd EA, Innes N, Clarkson J. Complete or ultraconservative removal of decayed tissue in unfilled teeth. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD003808. doi: 10.1002/14651858.CD003808.pub2. PMID 16856019
- [Background] JOE Editorial Board. Treatment of the primary tooth: an online study guide. J Endod. 2008 May;34(5 Suppl):e107-10. doi: 10.1016/j.joen.2007.08.004. PMID 18457686
- [Background] Garber AM, Phelps CE. Economic foundations of cost-effectiveness analysis. J Health Econ. 1997 Feb;16(1):1-31. doi: 10.1016/s0167-6296(96)00506-1. PMID 10167341
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Martins-Junior PA, Ramos-Jorge J, Paiva SM, Marques LS, Ramos-Jorge ML. Validations of the Brazilian version of the Early Childhood Oral Health Impact Scale (ECOHIS). Cad Saude Publica. 2012 Feb;28(2):367-74. doi: 10.1590/s0102-311x2012000200015. PMID 22331162
- [Result] Floriano I, Bonini GC, Matos R, Novaes TF, Ekstrand KR, Mendes FM, Braga MM. How different do visuo-tactile criteria assess caries lesions activity status on occlusal surfaces? Oral Dis. 2015 Apr;21(3):299-307. doi: 10.1111/odi.12265. Epub 2014 Aug 14. PMID 24912618